CLINICAL TRIAL: NCT01240590
Title: A Phase I/II Trial of Crolibulin (EPC2407) Plus Cisplatin in Adults With Solid Tumors With a Focus on Anaplastic Thyroid Cancer (ATC)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, James Gulley, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 110027; 11-C-0027
Record Dates: First submitted 2010-11-11; First posted 2010-11-15 (Estimated); Results first posted 2015-12-31 (Estimated); Last update posted 2017-04-10 (Actual); Status verified 2017-02

CONDITIONS: Solid Tumor; Anaplastic Thyroid Cancer
Keywords: Anaplastic Thyroid Cancer; Crolibulin; Solid Tumors; ATC
MeSH Terms: conditions — Thyroid Carcinoma, Anaplastic | interventions — crolibulin; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Ph I Level -1: Cisplatin + Crolibulin (Experimental): 75mg/m(2) Cisplatin + 8 mg/m(2) Crolibulin
  Interventions: Drug: Crolibulin; Drug: Cisplatin
- Ph I Level 1: Cisplatin + Crolibulin (Active Comparator): 75mg/m(2) Cisplatin + 13 mg/m(2) Crolibulin
  Interventions: Drug: Crolibulin; Drug: Cisplatin
- Ph I Level 2: Cisplatin + Crolibulin (Active Comparator): 100mg/m(2) Cisplatin + 13 mg/m(2) Crolibulin
  Interventions: Drug: Crolibulin; Drug: Cisplatin
- Ph II Level 3: Cisplatin + Crolibulin (Active Comparator): 100mg/m(2) Cisplatin + 20 mg/m(2) Crolibulin
  Interventions: Drug: Crolibulin; Drug: Cisplatin
- Ph II Level 4: Cisplatin (Active Comparator): 100mg/m(2) Cisplatin
  Interventions: Drug: Cisplatin

INTERVENTIONS:
Drug: Crolibulin — Phase I:Dose Level (DL) 1 - 13 mg/m(2) intravenous (IV),DL 2 - 13 mg/m(2) IV, DL 3 - 20 mg/m(2) IV. Phase II: 20 mg/m(2)
  Other Names: EPC2407
  Arms: Ph I Level -1: Cisplatin + Crolibulin; Ph I Level 1: Cisplatin + Crolibulin; Ph I Level 2: Cisplatin + Crolibulin; Ph II Level 3: Cisplatin + Crolibulin
Drug: Cisplatin — Phase I:Dose Level (DL) 1- 75 mg/m(2) intravenous (IV),DL 2 - 100 mg/m(2),DL 3 - 100 mg/m(2). Phase II: 100 mg/m(2)
  Other Names: CDDP

SUMMARY:
Background:

Anaplastic thyroid cancer (ATC) is one of the most aggressive of all solid tumors; chemotherapy and surgery have had no impact on local control or survival of patients, with a median survival of 3-7 months.

Crolibulin (EPC2407) is a microtubulin inhibitor that has been shown to have direct antitumor effects in vivo and in vitro, destabilizing spindles and inducing apoptosis, resulting in the disruption of neovascular endothelial cells with disruption of blood flow to the tumor. Early clinical studies with combretastatin, from which crolibulin is derived, demonstrated efficacy in a subset of patients with ATC.

Objectives:

The primary objective in the Phase I portion is to assess the safety and tolerability of cisplatin and crolibulin given in a 21-day cycle in dose-seeking cohorts.

We will assess the toxicities of crolibulin coadministered with cisplatin, evaluate dose-limiting toxicities (DLTs) and determine the maximum tolerated dose (MTD) for the combination.

The primary objective in the Phase II portion is to compare the combination crolibulin plus cisplatin versus cisplatin alone in adults with ATC by assessing the duration of progression-free survival (PFS); comparison of the response rates as evaluated by Response Evaluation Criteria in Solid Tumors (RECIST) will be an important secondary objective.

We plan on biochemical and immunohistochemical analysis of several tumor parameters including mitotic index, expression of several proteins including epidermal growth factor receptor (EGFR), vascular endothelial growth factor receptor (VEGFR), BRAF, excision repair cross-complementation group 1 (ERCC1) and tumor protein p53 (TP53). Where sufficient tissue is available we will also perform gene expression analysis, micro ribonucleic acid (microRNA) array analysis, and compare these with 3-deoxy-3 -[(18)F] fluorothymidine (FLT)-positron emission tomography (PET) and tumor growth rate constant.

Eligibility:

Phase I: adults age 18 and older with unresectable, recurrent or metastatic solid tumors.

Phase II: adults age 18 and older with anaplastic thyroid cancer.

In the phase II portion disease must be evaluable by RECIST.

All patients must have adequate hepatic, renal, and bone marrow function.

Design:

The Phase I component consists of dose-escalation cohorts of three to six patients, in which all patients receive both the study drug crolibulin with cisplatin. The MTD and DLT will be determined based on toxicities during the first three weeks of combined therapy.

The Phase II component will be a randomization study, to either crolibulin with cisplatin or cisplatin monotherapy. Patients randomized to cisplatin alone will have the opportunity the opportunity to cross over to the crolibulin arm in the event of tumor progression.

Drug administration will take place on days 1, 2, and 3 for crolibulin, and on day 1 for cisplatin, on a 21-day cycle.

Maximum number of patients for planned enrollment is 70. During the Phase I portion of the study, dose-seeking cohorts of three to six patients will be enrolled until MTD / DLT is reached for a maximum of three dose cohorts [up to 24 patients if one assumes an expansion cohort to twelve patients at the recommended phase 2 (RP2) dose]. During the randomized Phase II trial comparing the activity of the combination of crolibulin plus cisplatin with cisplatin alone it is estimated that a maximum of 40 patients will be enrolled [1:1 randomization 20 + 20 = 40 patients], and we will allow for 6 extra patients to be enrolled to compensate for a small number of non-evaluable patients.

DETAILED DESCRIPTION:
Background:

Anaplastic thyroid cancer (ATC) is one of the most aggressive of all solid tumors; chemotherapy and surgery have had no impact on local control or survival of patients, with a median survival of 3-7 months.

Crolibulin (EPC2407) is a microtubulin inhibitor that has been shown to have direct antitumor effects in vivo and in vitro, destabilizing spindles and inducing apoptosis, resulting in the disruption of neovascular endothelial cells with disruption of blood flow to the tumor.

Objectives:

The primary objective in the Phase I portion is to assess the safety and tolerability of cisplatin and crolibulin given in a 21-day cycle in dose-seeking cohorts.

We will assess the toxicities of crolibulin coadministered with cisplatin, evaluate dose-limiting toxicities (DLTs) and determine the maximum tolerated dose (MTD) for the combination.

The primary objective in the Phase II portion is to compare the combination crolibulin plus cisplatin versus cisplatin alone in adults with ATC by assessing the duration of progression-free survival (PFS); comparison of the response rates as evaluated by Response Evaluation Criteria in Solid Tumors (RECIST) will be an important secondary objective.

We plan on biochemical and immunohistochemical analysis of several tumor parameters including mitotic index, expression of several proteins including epidermal growth factor receptor (EGFR), vascular endothelial growth factor receptor (VEGFR), BRAF, ERCC1 and tumor protein p53 (TP53). Where sufficient tissue is available we will also perform gene expression analysis, microRNA array analysis, and compare these with 3-deoxy-3-[(18)F] fluorothymidine (FLT)-positron emission tomography (PET) and tumor growth rate constant.

Eligibility:

Phase I: adults age 18 and older with unresectable, recurrent or metastatic solid tumors.

Phase II: adults age 18 and older with anaplastic thyroid cancer.

In the phase II portion disease must be evaluable by RECIST.

All patients must have adequate hepatic, renal, and bone marrow function.

Design:

The Phase I component consists of dose-escalation cohorts of three to six patients, in which all patients receive both the study drug crolibulin with cisplatin. The MTD and DLT will be determined based on toxicities during the first three weeks of combined therapy. After a minimum of four cycles of concurrent cisplatin and crolibulin, if the patient is achieving clinical benefit in the opinion of the investigator but can no longer tolerate cisplatin, the patient may receive crolibulin alone until he or she experiences unacceptable toxicity or progressive disease.

The Phase II component will be a randomization study, to either crolibulin with cisplatin or cisplatin monotherapy. Patients randomized to cisplatin alone will have the opportunity to cross over to the crolibulin arm in the event of tumor progression. After a minimum of four cycles of concurrent cisplatin and crolibulin, if the patient is achieving clinical benefit in the opinion of the investigator but can no longer tolerate cisplatin, the patient may receive crolibulin alone until he or she experiences unacceptable toxicity or progressive disease.

Drug administration will take place on days 1, 2, and 3 for crolibulin, and on day 1 for cisplatin, on a 21-day cycle.

Maximum number of patients for planned enrollment is 70. During the Phase I portion of the study, dose-seeking cohorts of three to six patients will be enrolled until MTD / DLT is reached for a maximum of three dose cohorts [up to 24 patients if one assumes an expansion cohort to twelve patients at the recommended phase 2 (RP2) dose]. During the randomized Phase II trial comparing the activity of the combination of crolibulin plus cisplatin with cisplatin alone it is estimated that a maximum of 40 patients will be enrolled [1:1 randomization 20 + 20 = 40 patients], and we will allow for 6 extra patients to be enrolled to compensate for a small number of non-evaluable patients.

ELIGIBILITY:
* INCLUSION CRITERIA:

Pathologic confirmation of cancer by the Laboratory of Pathology, National Cancer Institute (NCI)

Phase I: Diagnosis of recurrent, metastatic or primary unresectable solid tumor that does not have curative standard treatment.

Phase II: Diagnosis of recurrent, metastatic or primary unresectable anaplastic thyroid cancer (ATC), including ATC as part of a thyroid carcinoma of another histologic subtype.

Measurable disease at presentation with disease measurable by Response Evaluation Criteria in Solid Tumors (RECIST) required in the phase II cohort.

A life expectance of at least 3 months as evidenced by Eastern Cooperative Oncology Group (ECOG) performance status 0-1.

Age greater than or equal to 18 years

Last dose of chemotherapy or experimental therapy more than 4 weeks (6 weeks in the case of nitrosourea) prior to enrollment date; unless the last therapy consisted of an oral agent whose average half life is known to be less than 48 hours in which case only 2 weeks need to have elapsed. Regardless of the therapy, any toxicity greater than Common Terminology Criteria in Adverse Events (CTCAE) grade 1 from previous anti-cancer therapy must have been resolved.

Last radiotherapy treatment 4 weeks prior to starting treatment with this protocol with the exception of palliative radiotherapy and there must be sites of measurable disease that did not receive radiation.

* Organ and marrow function as defined:
* total bilirubin < 1.5 times the upper limit of reference range (ULRR), unless the patient meets the criteria for Gilbert's Syndrome
* alanine aminotransferase (ALT), aspartate aminotransferase (AST) and alkaline phosphatase (ALP) all three < 2.5 times the ULRR, or < 5 times the ULRR if judged by the investigator to be related to liver metastases
* serum creatinine ULRR or creatinine clearance greater than or equal to 50 mL/minute (calculated by Cockcroft-Gault formula or measured in a timed urine collection)
* serum calcium below the CTCAE grade 1 upper limit (11.5mg/dL or 2.9 mmol/L). In cases where the serum calcium is below the normal range, the calcium adjusted for albumin is calculated and substituted for the measured value.
* Serum potassium greater than the lower limit of normal (LLN) and < 5.5 mmol/L.
* Serum magnesium greater than the LLN and < 3.0 mg/dL or 1.23 mmol/L.
* absolute neutrophil count greater than or equal to 1000/mm(3)
* platelet count (Bullet) 100,000/m m(3)
* Prothrombin time (PT) less than or equal to 4 seconds above ULN and partial thromboplastin time (PTT) less than or equal to 10 seconds above ULN.

Ability to understand and sign an informed consent document.

Provision of informed consent prior to any study-related procedures

Negative pregnancy test for women of childbearing potential

Ability and willingness to follow the guidelines of the clinical protocol including visits to NCI, Bethesda, Maryland for treatment and follow up visits.

Because the effects of chemotherapy on the developing human fetus are potentially harmful, female patients must be one year post-menopausal, surgically sterile, or using an acceptable method of contraception during and continued after the last dose of study medications (oral contraceptives, barrier methods, approved contraceptive implant, long-term injectable contraception, intrauterine device or tubal ligation). Male patients must be surgically sterile or using an acceptable method of contraception during their participation in this study. Contraceptive use will continue for at least two months after the last dose of study medication.

EXCLUSION CRITERIA:

Patients with cancer potentially curable by surgical excision alone or patients who have not received therapy that might be considered standard and potentially curable.

Evidence of severe or uncontrolled systemic disease or any concurrent condition including, but not limited to symptomatic congestive heart failure, unstable angina pectoris, unstable hypertension, seizure disorder, or psychiatric illness which in the Investigators opinion makes it undesirable for the patient to participate in the trial or which would jeopardize compliance with the protocol.

Untreated brain metastases (or local treatment of brain metastases within the last three months) due to the poor prognosis of these patients and difficulty ascertaining the cause of neurologic toxicities.

During Phase II enrollment: Prior therapy with cisplatin. (Cisplatin will be allowed as prior therapy during Phase I enrollment.)

Women who are currently pregnant or breast-feeding, due to the possible adverse effects on the developing fetus and infant.

During Phase II enrollment: The presence of a second malignancy within the last 2 years, other than squamous cell carcinoma of the skin or in situ cervical cancer because it will complicate the primary objective of the study. Cancer survivors who have been free of disease for at least two years can be enrolled in this study.

Patients with evidence of a bleeding diathesis that cannot be corrected with standard therapy or factor replacement.

Any unresolved toxicity greater than CTCAE grade 1 (except alopecia, and certain other unresolved CTCAE Grade 2 toxicities including bone marrow hypocellularity, lymphopenia, infusion-related reaction, infusion site extravasation, injection site reaction, portal vein hypertension, obesity) from previous anti-cancer therapy. Patients with grade 1 neuropathy will be evaluated on a case by case basis for entry into study. Pre-chemotherapy medical conditions will be taken into consideration.

Major surgery with incompletely healed surgical incision before starting study therapy.

Clinically significant cardiovascular event (e.g. myocardial infarction, superior vena cava syndrome (SVC), New York Heart Association (NYHA) classification of heart disease greater than or equal to 2 (see Appendix C) within 3 months before entry; or presence of cardiac disease that, in the opinion of the Investigator, increases the risk of ventricular arrhythmia.

History of arrhythmia (multifocal premature ventricular contractions PVCs), bigeminy, trigeminy, ventricular tachycardia, or uncontrolled atrial fibrillation) which is symptomatic or requires treatment (CTCAE grade 3) or asymptomatic sustained ventricular tachycardia. Atrial fibrillation, controlled on medication is not excluded.

Patients with a left ventricular ejection fraction less than the institutional lower limit of normal.

History (within the last 6 months) or presence of stroke/cerebrovascular accident.

Corrected QT interval (QTc) prolongation with other medications. If the medication can be discontinued and an alternative medication started that does not cause QTc prolongation, the patient would be eligible. If no alternative medication is available and the medication can not be discontinued for medical reasons, then the patient would not be eligible.

Congenital long Q wave, T wave (QT) syndrome, or 1st degree relative with unexplained sudden death under 40 years of age.

Presence of left bundle branch block (LBBB).

QTc with Bazett's correction that is not measurable, or greater than or equal to 480 msec on screening electrocardiogram (ECG). (Note: If a patient has a QTc interval greater than or equal to 480 msec on screening ECG, the screen ECG may be repeated twice (at least 24 hours apart). The average QTc from the three screening ECGs must be < 480 msec in order for the patient to be eligible for the study). Patients who are receiving a drug that has a risk of QTc prolongation (see Appendix C of the protocol) are excluded if QTc is greater than or equal to 460 msec.

Concurrent medication that may cause QTc prolongation or induce Torsades de Pointes: Those medications in Group One of Appendix C of the protocol will not be allowed. Those medications in Group Two of Appendix C of the protocol will be allowed.

Crolibulin is a substrate of cytochrome P450 2C8 (CYP2C8), P450 2C9(CYP2C9), P450 2C19 (CYP2C19) and P450 3A4 (CYP3A4). Strong inducers and inhibitors of these enzymes will constitute concomitant medications that are prohibited during the study (See protocol for the complete list). These medications include but are not limited to: for CYP2C8, montelukast and trimethoprim, for CYP2C9, lovastatin and sertraline, for CYP2C19, fluoxetine, ketoconazole, pantoprazole, omeprazole, rabeprazole, and ticlopidine, for CYP3A4, itraconazole, clarithromycin, erythromycin, telithromycin, and verapamil.

Hypertension not controlled by medical therapy (systolic blood pressure greater than 150 mm Hg or diastolic blood pressure greater than 100 mm Hg).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2011-01-26 (Actual); Primary Completion 2015-08-31 (Actual); Study Completion 2016-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Gulley, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Davies L, Welch HG. Increasing incidence of thyroid cancer in the United States, 1973-2002. JAMA. 2006 May 10;295(18):2164-7. doi: 10.1001/jama.295.18.2164. PMID 16684987
- [Background] Burgess JR, Tucker P. Incidence trends for papillary thyroid carcinoma and their correlation with thyroid surgery and thyroid fine-needle aspirate cytology. Thyroid. 2006 Jan;16(1):47-53. doi: 10.1089/thy.2006.16.47. PMID 16487013
- [Background] Truong T, Rougier Y, Dubourdieu D, Guihenneuc-Jouyaux C, Orsi L, Hemon D, Guenel P. Time trends and geographic variations for thyroid cancer in New Caledonia, a very high incidence area (1985-1999). Eur J Cancer Prev. 2007 Feb;16(1):62-70. doi: 10.1097/01.cej.0000236244.32995.e1. PMID 17220706
- [Derived] Cabanillas ME, McFadden DG, Durante C. Thyroid cancer. Lancet. 2016 Dec 3;388(10061):2783-2795. doi: 10.1016/S0140-6736(16)30172-6. Epub 2016 May 27. PMID 27240885
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2011-C-0027.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The phase II portion was not completed because it was impossible to recruit.
Groups:
- Level -1: Cisplatin + Crolibulin: 75mg/m(2) Cisplatin + 8 mg/m(2) Crolibulin Drug: Crolibulin Phase I:Dose Level (DL) 1 - 13 mg/m(2) intravenous (IV),DL 2 - 13 mg/m(2) IV, DL 3 - 20 mg/m(2) IV. Phase II: 20 mg/m(2) Drug: Cisplatin Phase I:Dose Level (DL) 1- 75 mg/m(2) intravenous (IV),DL 2 - 100 mg/m(2),DL 3 - 100 mg/m(2). Phase II: 100 mg/m(2)
- Level 1: Cisplatin + Crolibulin: 75mg/m(2) Cisplatin + 13 mg/m(2) Crolibulin Drug: Crolibulin Phase I:Dose Level (DL) 1 - 13 mg/m(2) intravenous (IV),DL 2 - 13 mg/m(2) IV, DL 3 - 20 mg/m(2) IV. Phase II: 20 mg/m(2) Drug: Cisplatin Phase I:Dose Level (DL) 1- 75 mg/m(2) intravenous (IV),DL 2 - 100 mg/m(2),DL 3 - 100 mg/m(2). Phase II: 100 mg/m(2)
- Level 2: Cisplatin + Crolibulin: 100mg/m(2) Cisplatin + 13 mg/m(2) Crolibulin Drug: Crolibulin Phase I:Dose Level (DL) 1 - 13 mg/m(2) intravenous (IV),DL 2 - 13 mg/m(2) IV, DL 3 - 20 mg/m(2) IV. Phase II: 20 mg/m(2) Drug: Cisplatin Phase I:Dose Level (DL) 1- 75 mg/m(2) intravenous (IV),DL 2 - 100 mg/m(2),DL 3 - 100 mg/m(2). Phase II: 100 mg/m(2)
- Level 3: Cisplatin + Crolibulin: 100mg/m(2) Cisplatin + 20 mg/m(2) Crolibulin Drug: Crolibulin Phase I:Dose Level (DL) 1 - 13 mg/m(2) intravenous (IV),DL 2 - 13 mg/m(2) IV, DL 3 - 20 mg/m(2) IV. Phase II: 20 mg/m(2) Drug: Cisplatin Phase I:Dose Level (DL) 1- 75 mg/m(2) intravenous (IV),DL 2 - 100 mg/m(2),DL 3 - 100 mg/m(2). Phase II: 100 mg/m(2)
- Level 4: Cisplatin: 100mg/m(2) Cisplatin Drug: Cisplatin Phase I:Dose Level (DL) 1- 75 mg/m(2) intravenous (IV),DL 2 - 100 mg/m(2),DL 3 - 100 mg/m(2). Phase II: 100 mg/m(2)
Period: Phase I
Arm/Group | Level -1: Cisplatin + Crolibulin | Level 1: Cisplatin + Crolibulin | Level 2: Cisplatin + Crolibulin | Level 3: Cisplatin + Crolibulin | Level 4: Cisplatin
Started | 0 | 6 | 3 | 0 | 0
Completed | 0 | 6 | 0 | 0 | 0
Not Completed | 0 | 0 | 3 | 0 | 0
Not completed — Refused further treatment | 0 | 0 | 3 | 0 | 0
Period: Phase II
Arm/Group | Level -1: Cisplatin + Crolibulin | Level 1: Cisplatin + Crolibulin | Level 2: Cisplatin + Crolibulin | Level 3: Cisplatin + Crolibulin | Level 4: Cisplatin
Started | 0 | 0 | 0 | 17 | 1
Completed | 0 | 0 | 0 | 15 | 0
Not Completed | 0 | 0 | 0 | 2 | 1
Not completed — Refused further treatment | 0 | 0 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ph I Level -1: Cisplatin + Crolibulin | Ph I Level 1: Cisplatin + Crolibulin | Ph I Level 2: Cisplatin + Crolibulin | Ph II Level 3: Cisplatin + Crolibulin | Ph II Level 4: Cisplatin | Total
Number analyzed (Participants) | 0 | 6 | 3 | 17 | 1 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years |  | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years |  | 2 | 3 | 12 | 0 | 17
  >=65 years |  | 4 | 0 | 5 | 1 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] |  | 68.03 (8.09) | 51.53 (7.45) | 58.76 (8.44) | 70.3 (0) | 60.45 (9.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 1 | 1 | 4 | 1 | 7
  Male |  | 5 | 2 | 13 | 0 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino |  | 1 | 0 | 1 | 0 | 2
  Not Hispanic or Latino |  | 5 | 3 | 16 | 1 | 25
  Unknown or Not Reported |  | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  | 0 | 0 | 0 | 0 | 0
  Asian |  | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander |  | 0 | 0 | 0 | 0 | 0
  Black or African American |  | 0 | 0 | 0 | 0 | 0
  White |  | 5 | 3 | 17 | 0 | 25
  More than one race |  | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported |  | 1 | 0 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States |  | 6 | 3 | 17 | 1 | 27

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Cisplatin (Phase I)
Description: MTD is defined as the dose level immediately preceding the dose level at which 2 dose limiting toxicities (DLT) occurred. A DLT is defined as a hematologic or non-hematologic adverse event judged to be possibly, probably, or definitely related to cisplatin per the Common Terminology Criteria in Adverse Events (CTCAE).
Time Frame: 3 weeks
Measure: Number; unit: mg/m^2
Groups:
- All Participants: All participants who received at least one dose of 75-100 mg/m(2) cisplatin intravenously.
Arm/Group | All Participants
Number analyzed (Participants) | 9
mg/m^2 | 100

2. Primary Outcome: Maximum Tolerated Dose (MTD) of Crolibulin (Phase I)
Description: as for outcome 1
Time Frame: 3 weeks
Measure: Number; unit: mg/m^2
Groups:
- All Participants: All participants who received at least one dose of 8-20 mg/m(2)crolibulin intravenously.
Arm/Group | All Participants
Number analyzed (Participants) | 9
mg/m^2 | 20

3. Primary Outcome: Progression Free Survival (Phase II)
Description: Progression free survival (PFS) is defined as the duration of time from start of study treatment to time of progression. Response is determined by the Response Evaluation Criteria in Solid Tumors (RECIST) and is defined as: Complete Response (CR) is disappearance of all target lesions; Partial Response (PR) is at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD. Progressive disease (PD) is at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions; and stable disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.
Time Frame: 6 weeks
Population: The outcome was not met because the patients died and were not scanned before their death.
Arm/Group | Ph II Level 3: Cisplatin + Crolibulin | Ph II Level 4: Cisplatin
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Number of Participants With Serious and Non-Serious Adverse Events (Phase I & II)
Description: Here is the number of participants with serious and non-serious adverse events. For a detailed list of adverse events, see the adverse event module.
Time Frame: 4 years, 6 months and 26 days
Measure: Number; unit: participants
Arm/Group | Ph I Level -1: Cisplatin + Crolibulin | Ph I Level 1: Cisplatin + Crolibulin | Ph I Level 2: Cisplatin + Crolibulin | Ph II Level 3: Cisplatin + Crolibulin | Ph II Level 4: Cisplatin
Number analyzed (Participants) | 0 | 6 | 3 | 17 | 1
participants |  | 6 | 1 | 16 | 1

5. Secondary Outcome: Number of Participants Who Underwent Medically-Necessary Interventions
Description: Enrolled participants who had surgical procedures deemed medically necessary for their clinical care.
Time Frame: 4.5 years
Measure: Count of Participants; unit: Participants
Groups:
- Ph I Level: -1 Cisplatin & Crolibulin: 75 mg/m(2) Cisplatin + 8 mg/m(2) Crolibulin
- Ph I Level: 1 Cisplatin & Crolibulin: 75 mg/m(2) Cisplatin + 13 mg/m(2) Crolibulin
- Ph I Level: 2 Cisplatin & Crolibulin: 100 mg/m(2) Cisplatin + 13 mg/m(2) Crolibulin
- Ph II Level: 3 Cisplatin & Crolibulin: 100 mg/m(2) Cisplatin + 20 mg/m(2) Crolibulin
- Ph II Level: 4 Cisplatin: 100 mg/m(2) Cisplatin
Arm/Group | Ph I Level: -1 Cisplatin & Crolibulin | Ph I Level: 1 Cisplatin & Crolibulin | Ph I Level: 2 Cisplatin & Crolibulin | Ph II Level: 3 Cisplatin & Crolibulin | Ph II Level: 4 Cisplatin
Number analyzed (Participants) | 0 | 6 | 3 | 17 | 1
Participants
  Gastrostomy | 0 | 1 | 0 | 0 | 0
  Trachesostomy | 0 | 0 | 0 | 1 | 0
  Cholecystectomy | 0 | 0 | 0 | 1 | 0
  No medically-necessary procedures | 0 | 5 | 3 | 15 | 1

6. Secondary Outcome: Tumor Growth Rate Constant
Description: Difference in time (days) required for the treated tumors to reach a predetermined target size.
Time Frame: 21 days
Population: This outcome measure was not analyzed because few if any re-assessments were done, thus there was not enough data to assess the growth rate constant on the patients.
Arm/Group | Ph I Level -1: Cisplatin + Crolibulin | Ph I Level 1: Cisplatin + Crolibulin | Ph I Level 2: Cisplatin + Crolibulin | Ph II Level 3: Cisplatin + Crolibulin | Ph II Level 4: Cisplatin
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 4 years, 6 months and 26 days
Arm/Group | Ph I Level: -1 Cisplatin & Crolibulin | Ph I Level: 1 Cisplatin & Crolibulin | Ph I Level: 2 Cisplatin & Crolibulin | Ph II Level: 3 Cisplatin & Crolibulin | Ph II Level: 4 Cisplatin
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/6 | 0/3 | 0/17 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/0 | 1/6 | 0/3 | 5/17 | 1/1
Other Adverse Events (participants affected / at risk) | 0/0 | 6/6 | 1/3 | 16/17 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ph I Level: -1 Cisplatin & Crolibulin (N=0) | Ph I Level: 1 Cisplatin & Crolibulin (N=6) | Ph I Level: 2 Cisplatin & Crolibulin (N=3) | Ph II Level: 3 Cisplatin & Crolibulin (N=17) | Ph II Level: 4 Cisplatin (N=1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neck edema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ph I Level: -1 Cisplatin & Crolibulin (N=0) | Ph I Level: 1 Cisplatin & Crolibulin (N=6) | Ph I Level: 2 Cisplatin & Crolibulin (N=3) | Ph II Level: 3 Cisplatin & Crolibulin (N=17) | Ph II Level: 4 Cisplatin (N=1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 6 (7) | 0 (0)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Alkalosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 3 (5) | 0 (0) | 11 (52) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 7 (8) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac troponin I increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 8 (37) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 10 (33) | 0 (0)
Fatigue (General disorders) | 0 (0) | 2 (4) | 0 (0) | 3 (3) | 0 (0)
Fever (General disorders) | 0 (0) | 2 (3) | 0 (0) | 3 (3) | 0 (0)
Flu like symptoms (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
General disorders and administration site conditions-Other, specify (General disorders) | 0 | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Mild left neck discomfort
GGT increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
hemoglobinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 1 (1) | 1 (2) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 3 (3) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (4) | 0 (0) | 3 (8) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 10 (68) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (7) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 2 (5) | 1 (1) | 9 (16) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 3 (4) | 1 (1) | 8 (17) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 4 (5) | 1 (1) | 11 (22) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (4) | 0 (0)
Infections and infestations - Other, specify (Oral thrush) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion site extravasation (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 3 (9) | 0 (0) | 9 (28) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metabolism and nutrition disorders - Other, specify (Amylase) (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (4) | 0 (0) | 7 (12) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (5) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 2 (4) | 1 (1) | 9 (21) | 0 (0)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (4) | 0 (0)
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0)
Weight loss (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 0 (0) | 2 (3) | 0 (0) | 2 (3) | 0 (0)

LIMITATIONS AND CAVEATS:
The phase II portion was not completed because it was impossible to recruit.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No